CLINICAL TRIAL: NCT01947400
Title: Does Use of the AIDET (Acknowledge, Introduce, Duration, Explanation, Thank) Method for Physician-patient Communication Improve Patient Satisfaction in a Real World Setting as Measured by Modified HCAHPS (Hospital Consumer Assessment of Health Plans Survey) Scores?
Brief Title: Effect of AIDET on Physician-Patient Communication
Acronym: AIDET
Status: Terminated | Type: Observational
Why Stopped: The data that was critical to the study was not able to be obtained.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201200279
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Physician Communication
Keywords: Physician and Patient Communication; Acknowledge Introduce Duration Explanation Thank; Hospital Consumer Assessment of Health Plans Survey
MeSH Terms: interventions — Hospitalists

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalists: AIDET Training
  Interventions: Other: Hospitalists

INTERVENTIONS:
Other: Hospitalists — AIDET Training

SUMMARY:
Patient satisfaction is an important aspect of care and is gaining increasing importance as a measure of Healthcare quality. Tools for improving physician-patient communication are available but have not yet been tested in the Hospital setting. The purpose of this project is to determine if training in AIDET (Acknowledge, Introduce, Duration, Explanation, Thank) communication method improves physician-patient communication. Patient satisfaction data will be compared to historical controls using modified HCAHPS (Hospital Consumer Assessment of Health Plans Survey) as the primary outcome measure. In addition, a validation of delivery of AIDET communication will be accomplished through administration of questionnaires to patients.

DETAILED DESCRIPTION:
This is a process of change study, which will compare HCAHPS patient satisfaction surveys before and after the Hospitalist receives AIDET physician-patient communication training. Once the Hospitalists agree to participate in the study, they will receive AIDET training by a Studor Group certified trainer. Both before and after the training intervention, Hospitalists' use of the AIDET method will be validated by having patients complete anonymous questionnaires during their hospital stay.

All HCAHPS surveys will be conducted by an external patient satisfaction survey vendor, and information will be de-identified both in terms of patient and specific Hospitalist. Validation questionnaires will be distributed by administrative staff, and will also be de-identified both in terms of patient and specific Hospitalist.

ELIGIBILITY:
Inclusion Criteria:

* Physicians: All physicians of the Hospital Medicine Service will be invited to participate

Exclusion Criteria:

* Any invited physicians who refuse to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians: Physicians of the Hospital Medicine Service
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
HCAHPS (Hospital Consumer Assessment of Health Plans Survey) Patient Satisfaction Scores | 1 year
AIDET Use Validation via Patient Questionnaires | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nila Radhakrishnan, MD, Principal Investigator — University of Florida; Robert Leverence, MD, Study Chair — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States